CLINICAL TRIAL: NCT01602107
Title: Optimizing Treatment Outcomes for Women With Stress Urinary Incontinence Through the Identification of Factors Contributing to Successful Interventions
Brief Title: The Effect of Pre-operative Pelvic Floor Muscle Exercise on Surgical Outcomes in Women With Stress Urinary Incontinence
Acronym: SUIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REH-503-11
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress; Urinary; Incontinence; Pelvic; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Participants in the control group will not receive therapist-supervised intervention. An exercise sheet briefly describing pelvic floor muscle exercises will be provided, as would be the standard practice from most physicians.
- Pelvic Floor Therapy (Experimental): Participants in the experimental group undergo and assessment and treatment by a registered physiotherapist. Treatments will include two sessions of biofeedback training, therapist-assisted strengthening exercises, and will a prescribed home exercise program to strengthen their pelvic floor muscles.
  Interventions: Other: Pelvic Floor muscle strengthening exercises

INTERVENTIONS:
Other: Pelvic Floor muscle strengthening exercises — Participants will attend regular physical therapy visits (weekly X 2 weeks, bi-weekly X 4 weeks, and continuing monthly) until the time of their surgery. they will then see the physical therapist for assessment, exercise and advice at 2 and 4 weeks after their surgery. During physical therapy visits, patients will receive two sessions of biofeedback training, and at each visit will work on strength and motor control exercises for their pelvic floor muscles.
  Other Names: Physical Therapy
  Arms: Pelvic Floor Therapy

SUMMARY:
Urinary incontinence (UI) affects up to 50% of adult populations and stress urinary incontinence (SUI) is the most common form of UI, accounting for approximately 60% of patients. Women are affected by SUI much more often than men. Urine leakage in women with SUI occurs on exertion or during tasks that increase pressure on the bladder such as sneezing or coughing. SUI has been shown to be a barrier to physical activity in women, and as such can contribute to the development of diseases and disorders associated with inactivity.

SUI appears to have many contributing factors such as structural damage (eg. tears in the pelvic organ supporting tissues), muscle weakness related to nerve injury or aging, or thinning of the urethral wall and/or its surrounding muscular sphincters. Currently the most common treatments for SUI are conservative therapy, which normally takes the form of exercise therapy provided by specialized nurses or physical therapists, and surgery, which is aimed at enhancing urethral support. Exercise therapy is effective, resulting in complete cure in 50% of cases, and surgery is effective for approximately 80% of patients but carries risks such as the development of urinary retention. It is currently not clear which treatment approach is better for which women.

Through the proposed research, the investigators aim to determine how to predict which patients will improve or be cured with exercise therapy such that surgery can be avoided. Specifically the investigators will determine what is different between patients in whom exercise therapy succeeds and in whom exercise therapy fails. The investigators will also determine whether physiotherapist-supervised training of the pelvic floor muscles before surgery improves surgical outcomes. The proposed research will enable us to better understand the female continence system and how it responds to physiotherapeutic intervention. It will help us to develop improved assessment procedures that can streamline patient management.

DETAILED DESCRIPTION:
It is hypothesized that participants in the physical therapy group will demonstrate greater improvements in pelvic floor muscle (PFM) function after treatment when compared to the control group. It is also expected that women in the physical therapy group will show better post-surgical outcomes when compared to the control group. The investigators will also develop and test a predictive model to identify those women with SUI who will benefit from physical therapy.

Objective 1: to evaluate characteristics predictive of the success or failure of PFM training in women with SUI.

To meet this objective, a cohort study will be used. Women with SUI will be recruited prospectively, will provide demographic information, will undergo a clinical evaluation of their PFM strength, will fill out the International Consultation on Incontinence Questionnaires (ICIQs), and will undergo an extensive evaluation of their continence system using ultrasound imaging. Ultrasound imaging will be used to measure muscle morphology (the presence and extent of PFM defect, PFM cross sectional area, urethral sphincter cross sectional area), fascial support (position of the bladder neck at rest and on Valsalva maneuver) and urethral mobility (amount of excursion of the urethra on coughing). A predictive multivariate binary logistic regression model will be developed to determine whether demographic variables, PFM strength, PFM morphology measures, fascial support or urethral mobility measured prior to the intervention can predict which women with SUI are cured after a standardized 12-week physical therapy program aimed at improving the strength, power, endurance and motor control of the PFMs.

Objective 2: to determine whether a program of pre- and peri-operative physical therapy aimed at improving the strength and motor control of the PFMs improves surgical outcomes relative to usual care in women with predominant symptoms of SUI.

Women who are waiting for surgery to treat symptoms of SUI at two hospital sites will be randomized to either a physical therapy group or a control group. Women assigned to the physical therapy group will receive a standardized 12 week program of PFM training prior to their surgery, will continue with these exercises until they undergo surgery, and will resume their exercises after surgery. The control group will receive usual care, which is a handout describing PFM exercises. The primary outcome of this study will be reported scores on patient-oriented ICIQs, which will be completed on entering the study, twelve weeks later, and at surgical follow up visit 12 weeks after surgery. Analysis of variance models will be used to compare outcomes between the physiotherapy group and the control group both before surgery and at 12 weeks after surgery. Chi Square models will assess whether cure rates are higher in women belonging to the physical therapy as compared to the control group.

Taken together, the results will direct clinical decision making around the delivery of appropriate interventions for women with SUI, particularly physical therapy and TVTand TVT-O surgery.

DESCRIPTION OF METHODS AND PROCEDURES

a) Study Design and Methodology: Subjects and Screening All women above the age of 18 who report symptoms of SUI and who have been evaluated by a urogynaecologist (Dr. M.A.Harvey or Dr. S. Johnston) at Kingston General Hospital (KGH), (Dr. K. Baker) at the Ottawa Hospital, (Dr. Magali Robert) at the Foothills Hospital in Calgary or (Dr. V. della Zazzera) at the Montfort Hospital in Ottawa and who have been deemed appropriate for TVT or TVT-O surgery and have decided to pursue this option will be asked by their physician if they are willing to be contacted by the investigators. For those who agree, they will receive a follow-up phone call to determine their interest in participating and, if appropriate, their eligibility. Eligible and interested participants will be instructed on how to complete a three-day bladder diary to record the number of daily episodes of urine leakage experienced over a typical three day period.

Volunteers will be scheduled to attend a baseline evaluation at the Pelvic Floor Laboratory at Queen's University or at the Dr. Linda McLean's Pelvic Floor Laboratory at the University of Ottawa. At this first visit, eligibility of the participant will be confirmed based on the bladder diary results (they must have experienced at least one episode of urine leakage over the three-day diary), a pad test and the absence of evidence of any neurological cause of pelvic floor muscle dysfunction.

Those who are still eligible will have their height and weight recorded, and bladder volume will be measured using trans-abdominal ultrasound (US) imaging. If the bladder volume is at least 250 ml, then the participant will begin a standardized pad test (i.e., a circuit of walking and stair climbing for 30 minutes, which has been shown to be highly sensitive and specific to the diagnosis of urinary incontinence. If the bladder volume is less than 250mL, the volunteer will be asked to drink 350mL of water and will wait until proper volume is attained. In this case, the volunteer will complete the study questionnaires described below while waiting for her bladder to fill. Once her bladder has been filled to 250mL, she will then begin the test. For the test, an incontinence pad will be weighed and adhered to her undergarment. The woman will then perform a standardized circuit of walking and stair climbing for 30 minutes, after which time the weight of the pad will be measured again. An increase in weight greater than 1g will confirm the presence of urine leakage and will confirm the participant's eligibility. If the participant is deemed ineligible at this point, she will be thanked for her participation and withdrawn from the remainder of the study.

At this point, volunteers who meet the bladder diary and pad test requirements will undergo an urogynecological screening exam by a research assistant.. This physical screening includes palpation to rule out pelvic mass(es), manual muscle testing to evaluate PFM strength, and sensory and reflex testing to rule out neurologic causes of incontinence. This will constitute the last step to evaluate participant's eligibility. If the participant has no evidence of pelvic mass or neurologic defects, all criteria are met, and the woman will enter the study.

At this same session, eligible participants will undergo a three-dimensional (3D) US imaging assessment of her pelvic region. Ultrasound imaging will be performed first in the lithotomy position using a transvaginal endoprobe to evaluate the urethral sphincter. Next, using a 3D curvilinear transducer, the PFMs will be visualized in the axial plane while the participant performs three repetitions of a maximal voluntary contraction. A 2D curvilinear transducer will then be used to capture video clips in the sagittal plane while the participant performs three repetitions of a Valsalva maneuver, and of a cough. The participant will then move to a standing position with a wide stance to allow for the curvilinear transducer to be applied against her perineum. She will be asked to repeat three repetitions of the Valsalva maneuver, and three repetitions of a maximal effort cough. This will conclude the US imaging testing section.

If they have not already been completed, the participant will conclude this session by completing the International Consultation on Incontinence Questionnaires (ICIQs) to evaluate their incontinence symptoms, and each participant will be given a standard educational sheet describing how to perform PFM strengthening exercises. They will be advised that they will be contacted to inform them whether they have been randomized to the physical therapy or control group. The entire baseline testing will take approximately 2.5 hours.

Randomization: Participants will be randomly assigned (1:1) to either the physical therapy group or the control group using a secure web-based computerized randomization system which will conceal future randomizations. Randomization will be stratified by site using permuted blocks of random size. Participant blinding is not possible in a study of this nature, however the research assistant performing the pre- and post-treatment assessments will remain blinded to group assignment during all data collection and processing.

Interventions: A total of 400 volunteers will be randomly assigned to each of the two experimental groups: Physical therapy or control group.

Physical Therapy Group The women in the standardized physical therapy treatment group will attend six sessions over a 12-week period. Treatments will be delivered by physical therapists with post-graduate training in urinary incontinence management. Physical therapists will have been trained on how to deliver the semi-standardized treatment protocol at their respective physical therapy clinics in the cities of Ottawa, Kingston or Calgary. In the first session, volunteers will learn to perform a proper PFM contraction using manual palpation and feedback to optimize PFM contraction quality in which they will learn to contract their PFMs before tasks that increase intra-abdominal pressure, such as coughing and postural perturbations (i.e., the Knack exercise). The women will be instructed to perform their prescribed exercises daily. At each 45-minute visit, the physical therapist will review and reinforce a proper PFM contraction technique, will evaluate PFM strength using a modified Oxford scale to provide feedback about progress, will review the Knack exercise (a quick contraction of the PFM during high intra-abdominal pressure) and will supervise the volunteer while she performs each task to ensure correct performance. The exercises will be progressed and compliance will be recorded as described below.

Control Group Participants in the control group will be asked to follow the recommendations on their pelvic floor muscle training educational sheet. They will be asked on follow up visits to report whether or not they attempted PFM exercises and if so, at what frequency.

Post-Intervention/Pre-surgical testing Women in both groups will return to the laboratory 12 weeks after the baseline testing described above. To ensure the evaluators remain blinded to group assignment, women will be asked not to reveal to the research assistant whether or not they received physical therapy treatment. The pre-surgical testing will repeat the baseline testing procedures in the same manner as described above (i.e., bladder diary, pad test, US imaging, questionnaires), with the exception that the neurological assessment that was initially used to determine eligibility will not be performed. After this pre-surgical testing, the women in the physical therapy group will be instructed to continue their exercise program and will visit their physical therapist every four weeks until their surgery. Women in the control group will be advised to continue their at-home PFM exercises, according to the information that was provided on their standard educational sheet.

Post-surgical intervention Only women in the physical therapy group will be advised to continue their exercise program starting the day after their TVT surgery. Each woman will visit her physical therapist one week, three weeks and five weeks after her surgery to ensure she is performing her PFM exercises correctly and to continue the progression of her PFM exercises according to her progress.

Post-surgical testing All women will return to the laboratory 12 weeks after their surgery and will be re-evaluated by the research assistant (still blinded to group assignment) using the ICIQs and the pad test. This post-surgical testing will last 45 minutes.

Long-term follow-up testing All women enrolled in the study will undergo long-term follow up using the bladder diary, ICIQs and pad test at 12 months and 2 years post-surgery. The ICIQs can be administered by phone, and this will be done by research assistants whenever patients cannot attend their follow-up visit(s) in order to reduce the number of participants lost to follow-up. This will conclude all participation and all women will be mailed or emailed a research study debriefing sheet outlining the study findings

ELIGIBILITY:
Inclusion Criteria:

* female
* minimum age of 18
* primary diagnosis of stress urinary incontinence by urogynaecologist
* on the surgical wait list for surgery to address stress urinary incontinence

Exclusion Criteria:

* currently pregnant or <6 months post-partum
* pelvic mass (es)
* pad test weight gain less than 1g at baseline testing
* no episode of SUI as demonstrated by a 3-day bladder diary
* having received more than 4 sessions of physical therapy in the past 5 years specifically for treating their symptoms of SUI
* detrusor instability as identified by routine urodynamics studies performed as part of the patient evaluation by the urogynaecologist
* prolapse (> POP-Q stage 2)
* are taking medications known to increase or alleviate incontinence
* not willing to cease other treatment for SUI treatment during the course of study
* fecal incontinence (e.g., pessary)
* prior urogynecological surgery to address urinary incontinence
* neurological impairments involving the central nervous system or the sacral nerves or known connective tissue disorders
* major psychiatric conditions which impact significantly with daily functioning and would prevent full participation in the study
* physical impairment that would prevent the participant from completing the 20-minute pad test (a major study outcome measure)
* in situ devices that would not be suitable for ultrasound testing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire: Female Lower Urinary Tract Symptoms (FLUTS) | 12 weeks before surgrey (TVT or TVT-O) to 12 weeks after surgery
  Changes in ICIQ FLUTS scores will be compared between treatment and control groups
Change in International Consultation on Incontinence Questionnaire - Short form score | 12 weeks before surgery (TVT or TVT-O) to 12 weeks after surgery
  Changes in questionnaire scores will be compared between treatment and control groups
Change in pad weight on a standardized 30 minute pad test | 12 weeks before surgery (TVT, TVT-O) to 12 weeks after surgery
  Change in pad weight (in g) on a standardized pad test will be compared between the treatment and control groups

SECONDARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire Quality of Life module score | 12 weeks before surgery (TVT, TVT-O) to 12 weeks after surgery
  Changes in ICIQ-FLUTS QoL scores will be compared between the treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, PhD, Principal Investigator — School Of Rehabilittion Therapy, Queen's University
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - School of Rehabilitation Therapy, Queen's University, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Montfort Hospital, Ottawa, Ontario

REFERENCES:
- [Derived] Antonio FI, Yamamoto G, Varette K, McLean L. One in four women with stress urinary incontinence who are taught "the knack" maneuver adopt this motor pattern while coughing: A prospective interventional cohort study. Neurourol Urodyn. 2023 Aug;42(6):1290-1298. doi: 10.1002/nau.25196. Epub 2023 May 2. PMID 37130076
- [Derived] McLean L, Charette M, Varette K, Brooks K, Harvey MA, Robert M, Baker K, Day A, Della Zazzera V, Sauerbrei E, Brison R. Pelvic floor muscle training as an adjunct to a midurethral sling: a single-blind randomised controlled trial. Int Urogynecol J. 2022 Apr;33(4):809-819. doi: 10.1007/s00192-020-04668-9. Epub 2021 Mar 3. PMID 33660001
- [Derived] Brooks KCL, Varette K, Harvey MA, Robert M, Brison RJ, Day A, Baker K, Della Zazzera V, Sauerbrei E, McLean L. A model identifying characteristics predictive of successful pelvic floor muscle training outcomes among women with stress urinary incontinence. Int Urogynecol J. 2021 Mar;32(3):719-728. doi: 10.1007/s00192-020-04583-z. Epub 2020 Nov 25. PMID 33237355